CLINICAL TRIAL: NCT03407378
Title: A Proof of Concept Study to Investigate the Effect of IPT803 Adjunct Treatment in Patients With Parkinson's Disease
Brief Title: A Study to Investigate a New Treatment in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tools4Patient (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: T1020-01
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessments ON regular PD treatment (Experimental): IPT803 Questionnaires Motor assessments on regular PD treatment Optional pharmacogenetic assessments Optional Blood-Oxygen-level Dependent Functional-MRI
  Interventions: Drug: IPT803; Genetic: Optional pharmacogenetic assessment; Other: Questionnaires; Other: Optional Blood-Oxygen-level Dependent functionalMRI; Other: Motor Assessments on regular PD treatment
- Assessments OFF regular PD treatment (Experimental): IPT803 Questionnaires Motor assessments before taking regular PD treatment Optional pharmacogenetic assessments Optional Blood-Oxygen-level Dependent Functional-MRI
  Interventions: Drug: IPT803; Genetic: Optional pharmacogenetic assessment; Other: Questionnaires; Other: Optional Blood-Oxygen-level Dependent functionalMRI; Other: Motor Assessments before taking regular PD treatment

INTERVENTIONS:
Drug: IPT803 — Administration of IPT803 three times a day for 12 weeks as add-on therapy to patient regular PD medication(s) or as a new therapy for drug naïve patients.
Genetic: Optional pharmacogenetic assessment — Blood sample of 3 milliliters for genotyping assessment (according to patient consent).
Other: Questionnaires — Personality, Health and Disease questionnaires completion during the study (Visits 1, 2, 3 and 4)
Other: Optional Blood-Oxygen-level Dependent functionalMRI — BOLD fMRI performed in a sub-group of patients, depending of randomization (exploratory)
Other: Motor Assessments before taking regular PD treatment — Regular PD treatment stopped 12 or 24 hours prior to Visits 2, 3 and 4 depending on the drug form (extended vs standard release). Motor assessments using UPDRS Part III are performed when patients are OFF regular PD treatment. Regular PD treatment is taken on site during the visit after the motor assessments are performed.
  Arms: Assessments OFF regular PD treatment
Other: Motor Assessments on regular PD treatment — Regular PD treatment is not modified before the visits. The motor assessments using UPDRS Part III are performed while the patient is on regular PD treatment.
  Arms: Assessments ON regular PD treatment

SUMMARY:
The purpose of this clinical trial conducted in patients with Parkinson's Disease is to study the relationship between patient individual profile and their response to IPT803 Adjunct Treatment (treatment response being characterized by movements improvement).

ELIGIBILITY:
Inclusion Criteria

1. Men or women of at least 35 years of age;
2. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures;
3. Have given written informed consent approved by the relevant Ethics Committee (EC)/Institutional Review Board (IRB) governing the study site(s);
4. Medically stable outpatients with idiopathic PD based on the MDS-PD criteria (Postuma et al 2015). The diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity or postural instability not caused by primary visual, vestibular, cerebellar, or proprioceptive dysfunction) being present, without any other known or suspected cause of Parkinson;
5. Patients with a Hoehn and Yahr Stage < 3;
6. Patients with a MMSE ≥ 26;
7. Patient stabilized with PD medication(s) e.g. levodopa, dopamine agonists, amantadine and/or Monoamine oxidase (MAO)-B inhibitors for at least 4 weeks prior to Visit 1 and and up to Visit 4 included or Drug naïve patients recently diagnosed with PD according to the criteria above and for whom PD medication(s) may be initiated after Visit 4;

   Exclusion Criteria
8. Pregnant (urine pregnancy test), breastfeeding, or willing to be pregnant during the study;
9. Presence of clinically significant medical or psychiatric condition that may increase the risk associated with study participation or investigational product/device administration or participation in any other type of medical research that may interfere with the interpretation of study results in the judgment of the sponsor/investigator or in an exclusion period according to national law, would make the subject inappropriate for entry into this study;
10. Has a history of psychotic symptoms requiring treatment with a neuroleptic medication within the past 12 months;
11. Any current primary psychiatric condition, including not stabilized mood disorders, personality disorders or mental retardation based on diagnostic following DSM-V;
12. Any known hypersensitivity to corn and/or corn-derived products;
13. Alcohol dependence or regular use of known drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and phencyclidine);
14. Any other relevant medical disorder/acute disease state judged by the Investigator as likely to interfere with study procedures or represent a risk for the patient;
15. Any close relationship with the investigators or employees or consultants of the sponsor (i.e. belonging to immediate family or subordination relationship);
16. Under legal protection, according to the national law (for French sites only);
17. Are persons who have previously received IPT803, have completed or withdrawn from this study or any other study investigating IPT803.
18. Change in the patient's regular PD medication(s) (dosage or dosing interval) or introduction of a new regular PD medication(s) within 4 weeks prior to Visit 1 and up to Visit 4 included;
19. Patients with motor complications (wearing off; dyskinesia) that would interfere with study procedures;
20. Patients with history or clinical features consistent with an atypical Parkinsonian syndrome (for example: supranuclear gaze palsy, clinically significant orthostatic hypotension);
21. History of surgical or invasive intervention for PD (pallidotomy, thalamotomy, deep brain stimulation, etc.);
22. Any Parkinson's disease-related feature or symptom that could interfere with the study conduct and results as assessed by the investigator.

    Exclusion Imaging (BOLD fMRI) criteria for patients following Imaging Procedure:
23. Patients unable to undergo MRI scans, including suffering from claustrophobia;
24. Have implanted or embedded metal objects or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field according to investigator site judgment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Patient's change from baseline of score as measured by Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS; Part III), after 12 weeks of IPT803 administration. | Time zero equals baseline equals (Visit 2 - Day 1 prior to IPT803 first dose) up to Visit 4 (Day 85)
  Part III of the MDS-UPDRS (or motor examination) assesses the motor abilities in PD patients at the time of the visit. This part measures 18 motor examinations such as speech, facial expression, tremor, rigidity, finger tapping, pronation-supination movements of hands, leg agility, arising from chair, gait.
  The qualified rater must score 34 items from 0 to 4, where 0 indicates a normal situation and 4 indicates that PD interferes severely in carrying out the task. The total score, being the sum of all these items, can be between 0 to 136.

SECONDARY OUTCOMES:
Patient's change from baseline of safety incidence as measured by the rate and severity of Treatment emergent adverse event (TEAEs). | Time zero equals baseline Visit 2 IPT803 first dose (Day 1) up to Visit 4 (Day 85)
Patient's change from baseline of motor and non-motor outcomes as measured by Part I, Part II and IV subscales of Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS). | From Visit 1 (Day -14 to Day -7) up to Visit 4 (Day 85)
  The MDS-UPDRS is divided into 4 parts. In each part, all items are rated on a scale from 0 (normal) to 4 (severe impairment).
  Part I assesses 15 items of non-motor aspects of experiences of daily living. Part IA is assessed by a qualified rater, Part IB is completed by the patient. The total score, being the sum of all these items, can be between 0 to 60.
  Part II comprises 13 items evaluating the impact of PD on patients' activities of daily living (ADL) over the week prior to the visit such as speech, salivation, swallowing, eating, handwriting, dressing, turning in bed, walking. It will be completed by the patient. The total score, being the sum of all these items, can be between 0 to 52.
  Part IV assesses motor complications of therapy, such as dyskinesias, motor fluctuations. This part (6 items) is completed by a qualified rater. The total score, being the sum of all these items, can be between 0 to 24.
The patient's change from baseline in disease severity as measured by the Parkinson's Disease Questionnaire (PDQ-39). | From Visit 2 (Day 1) up to Visit 4 (Day 85)
Patient's change from baseline of fatigue as measured by the Fatigue Severity Scale (FSS). | From Visit 1 (Day -14 to Day -7) up to Visit 4 (Day 85)
  The FSS is a self-administered questionnaire with 9 items assessing the severity of fatigue during the past 2 weeks. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement, where the addition of all numbers circled by patient get the final score.
Patient's change from baseline of sleep quality as measured by the Epworth Sleep Scale (ESS). | From Visit 1 (Day -14 to Day -7) up to Visit 4 (Day 85)
  The ESS assesses the overall level of daytime sleepiness. Eight items describe normative daily situations known to vary in their soporific qualities. Patients rate the likelihood of dozing off or falling asleep. The test is rated on a 4-point scale (0=would never doze off to 3=high chance of dozing off).
Investigator change from baseline in disease severity as measured by the Investigator Assessment of Changes (IGAC). | From Visit 2 (Day 1) up to Visit 4 (Day 85)
  IGAC is a subjective evaluation by the Investigator using a 0 to 10 Numeric Rating Scale (NRS) to answer the following question: "If you take into consideration all the various ways that motor control influences the patient and his/her life, how do you then evaluate the patient's motor condition today?", with 0 meaning "very bad" and 10 "very good".
Patient's change from baseline in disease severity as measured by the Patient Assessment of Changes (PGAC). | From Visit 2 (Day 1) up to Visit 4 (Day 85)
  PGAC is a subjective evaluation by the patient using a 0 to 10 Numeric Rating Scale (NRS) to answer the following question: "If you take into consideration all the various ways that motor control influences you and your life, how do you then evaluate your motor condition over the last week?", with 0 meaning "very bad" and 10 meaning "very good".
Patient's change from baseline above or equal to the minimal clinically important difference (MCID) of the motor score as measured by Part II and III subscales of Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS). | Time zero equals baseline (Visit 2 - Day 1 prior to IPT803 first dose) up to Visit 4 (Day 85)
  The Minimal Clinically Important Difference (MCID) is the smallest change in an outcome measure that is meaningful for patients.
  In the literature, the MCIDs of MDS-UPDRS Part II and Part III are respectively defined as a motor score reduction of 2 and 6 points. The motor scores are the sum of all items (ranging from 0-4) of each MDS-UPDRS subscale.
  Following endpoints will be measured:
  * A reduction above or equal to 2 points of MDS-UPDRS Part II motor score (minimum score= 0, maximal score= 52)
  * A reduction above or equal to 6 points of MDS-UPDRS Part III motor score (minimum score= 0, maximal score= 136)
  These endpoints will be interpreted as binary values: 0 (below) and 1 (above or equal).
Patient's change from baseline above or equal to 30 % or above or equal to 50 % of the motor score as measured by Part II and III subscales of MDS-UPDRS. | Time zero equals baseline (Visit 2 - Day 1 prior to IPT803 first dose) up to Visit 4 (Day 85)
  The motor scores are the sum of all items (ranging from 0-4) of each MDS-UPDRS subscale.
  Following endpoints will be measured:
  * A reduction above or equal to 30% of MDS-UPDRS Part II motor score
  * A reduction above or equal to 30% of MDS-UPDRS Part III motor score
  * A reduction above or equal to 50% of MDS-UPDRS Part II motor score
  * A reduction above or equal to 50% of MDS-UPDRS Part III motor score
  These endpoints will be interpreted as binary values: 0 (below) and 1 (above or equal).
Cronbach α assessment of MPsQ | at Visit 1 (Day -14 to Day -7), Visit 2 (Day 1) Visit 4 (Day 85)

OTHER OUTCOMES:
Patient's change from baseline of motor score, as measured by Inertial Measurement Unit (IMU) on Finger taping (FT) and Pronation-supination movement of the hands (PSH) during the 12-week treatment. | Time zero equals baseline equals (Visit 2 - Day 1 prior to IPT803 first dose) up to Visit 4 (Day 85)
  For all patients, objective quantitative movement will be collected with movement sensors (accelerometers and gyroscopes) during items 3.4 (FT) and 3.6 (PSH) of MDS-UPDRS Part III at Visits 2, 3 and 4.
  Collected data will be converted to continuous values on the same scale as MDS-UPDRS, from 0 to 4. The endpoint is defined as the patient's change from baseline of these continuous scales.
Patient's change from baseline of the regional brain activity as measured by BOLD fMRI measured by motor tasks performed during fMRI before and after single dose of IPT803. | On Day 1: prior to IPT 803 first dose and 60 minutes after IPT803 first dose
Patient's change of motor score, as measured by Part III subscale of MDS-UPDRS directly after IPT803 single dose. | On Day 1: prior to IPT 803 first dose and 30 minutes after IPT803 first dose
  The qualified rater must score 34 items from 0 to 4, where 0 indicates a normal situation and 4 indicates that PD interferes severely in carrying out the task. The total score, being the sum of all these items, can be between 0 to 136.

CONTACTS AND LOCATIONS:
Overall Officials: Pereira Alvaro, Study Director — Tools4Patient
Locations (10):
- United States (5):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Northwestern, Chicago, Illinois
  - Henry Ford, West Bloomfield, Michigan
  - Columbia, New York, New York
- CHU Liege - Liège University, Liège, Belgium
- France (4):
  - CHU Grenoble, Grenoble
  - CHU Poitiers, Poitiers
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU Purpan - Hopital Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No